CLINICAL TRIAL: NCT04198701
Title: Pulsed Field Ablation to Irreversibly Electroporate Tissue and Treat AF
Acronym: PULSED AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PULSED AF
Record Dates: First submitted 2019-12-10; First posted 2019-12-13 (Actual); Results first posted 2023-12-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: The study begins with a Pilot Phase, followed sequentially by a Pivotal Phase consisting of 3 arms enrolling simultaneously: Roll-in, Paroxysmal AF, Persistent AF
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Pilot (Experimental): First group of patients enrolled in the study.
  Interventions: Device: Medtronic PulseSelect Pulsed Field Ablation (PFA) System
- Pivotal - Roll-In (Experimental): First patient treated by each physician in the pivotal phase.
  Interventions: Device: Medtronic PulseSelect Pulsed Field Ablation (PFA) System
- Pivotal - Paroxysmal AF (Experimental): Non roll-in patients with paroxysmal AF (intermittent AF).
  Interventions: Device: Medtronic PulseSelect Pulsed Field Ablation (PFA) System
- Pivotal - Persistent AF (Experimental): Non roll-in patients with persistent AF (AF that lasts longer than 7 days).
  Interventions: Device: Medtronic PulseSelect Pulsed Field Ablation (PFA) System

INTERVENTIONS:
Device: Medtronic PulseSelect Pulsed Field Ablation (PFA) System — Adult subjects with a history of drug refractory recurrent symptomatic atrial fibrillation (AF) will undergo ablation of pulmonary veins and confirmation of entrance block and, where assessable, exit block with the PulseSelect PFA System.

SUMMARY:
The study is a prospective, multi-center, non-randomized, unblinded worldwide pre-market clinical study. The purpose of the study is to provide data demonstrating the safety and effectiveness of the PulseSelect™ PFA System for the treatment of atrial fibrillation (AF). The study will also provide first in human insights into clinical safety and device function of the PulseSelect PFA System for pulmonary vein isolation (PVI) as a treatment for AF. To this end, the clinical study has been designed into phases (Pilot and Pivotal), with each phase comprising a separate data set that will be analyzed and reported on per the below objectives.

ELIGIBILITY:
Inclusion Criteria:

1. Failure of at least one AAD (class I or III) for AF as evidenced by recurrent symptomatic AF, or intolerable side effects due to AAD.
2. A diagnosis of recurrent symptomatic paroxysmal or persistent AF:

   1. Symptomatic paroxysmal AF, which is defined as AF that terminates spontaneously or with intervention within 7 days of onset, documented by the following:

      1. physician's note indicating at least 2 symptomatic paroxysmal AF episodes occurring within 6 months prior to enrollment; and
      2. at least 1 ECG documented AF episode from any form of rhythm monitoring within 12 months prior to enrollment OR
   2. Symptomatic persistent AF, which is defined as continuous AF sustained beyond 7 days and less than 1 year, documented by the following:

      1. physician's note indicating at least 1 symptomatic persistent AF episode occurring within 6 months prior to enrollment; and
      2. any 24-hour continuous ECG recording documenting continuous AF within 6 months prior to enrollment; OR 2 ECGs from any form of rhythm monitoring taken at least 7 days apart, both showing continuous AF within 6 months prior to enrollment
3. Age 18 through 80 years old (or older than 18 if required by local law)

Exclusion Criteria:

1. Long-standing persistent AF (continuous AF that is sustained >12 months)
2. Left atrial diameter > 5.0 cm (anteroposterior)
3. Prior left atrial ablation or surgical procedure (including left atrial appendage closures)
4. Planned LAA closure procedure or implant of a permanent pacemaker, biventricular pacemaker, loop recorder/insertable cardiac monitor (ICM), or any type of implantable cardiac defibrillator (with or without biventricular pacing function) for any time during the follow-up period
5. Patient who is not on oral anticoagulation therapy for at least 3 weeks prior to the ablation procedure
6. Presence of a permanent pacemaker, biventricular pacemaker, loop recorder/insertable cardiac monitor (ICM), or any type of implantable cardiac defibrillator (with or without biventricular pacing function)
7. Presence of any pulmonary vein stents
8. Presence of any pre-existing pulmonary vein stenosis
9. Pre-existing hemidiaphragmatic paralysis
10. Presence of any cardiac valve prosthesis
11. Moderate to severe mitral valve stenosis
12. More than moderate mitral regurgitation (i.e., 3+ or 4+ MR)
13. Any cardiac surgery, myocardial infarction, PCI / PTCA or coronary artery stenting which occurred during the 3-month interval preceding the consent date
14. Unstable angina
15. NYHA Class III or IV congestive heart failure or documented left ventricular ejection fraction (LVEF) less than or equal to 35% measure by acceptable cardiac testing (e.g. TTE)
16. Primary pulmonary hypertension
17. Rheumatic heart disease
18. Thrombocytosis, thrombocytopenia
19. Any condition contraindicating chronic anticoagulation
20. Active systemic infection
21. Hypertrophic cardiomyopathy
22. Known reversible causes of AF, including but not limited to uncontrolled hyperthyroidism, severe untreated obstructive sleep apnea, and acute alcohol toxicity
23. Any cerebral ischemic event (strokes or TIAs) which occurred during the 6-month interval preceding the consent date
24. History of thromboembolic event within the past 6 months or evidence of intracardiac thrombus at the time of the procedure
25. Any woman known to be pregnant or breastfeeding, or any woman of childbearing potential who is not on a reliable form of birth regulation method or abstinence
26. Patient with life expectancy that makes it unlikely 12 months of follow-up will be completed
27. Current or anticipated participation in any other clinical trial of a drug, device or biologic during the duration of the study not pre-approved by Medtronic
28. Known allergies or hypersensitivities to adhesives
29. Unwilling or unable to comply fully with study procedures and follow-up
30. Unable to provide own informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Atul Verma, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (41):
- United States (27):
  - Grandview Medical Center, Birmingham, Alabama
  - Medical Center of the Rockies, Loveland, Colorado
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - BayCare Saint Joseph's Hospital, Tampa, Florida
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northwestern University Hospital, Chicago, Illinois
  - Iowa Heart Center, Des Moines, Iowa
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Southcoast Health System, Fall River, Massachusetts
  - Spectrum Health, Grand Rapids, Michigan
  - Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic (Rochester MN), Rochester, Minnesota
  - Saint Luke's Mid America Heart Institute, Kansas City, Missouri
  - The Valley Hospital, Ridgewood, New Jersey
  - Northwell Health - North Shore University Hospital, Manhasset, New York
  - NYU Langone Health - Heart Rhythm Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center- UPMC Presbyterian, Pittsburgh, Pennsylvania
  - St. David's Medical Center, Austin, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Swedish Medical Center Cherry Hill, Seattle, Washington
- John Hunter Hospital, New Lambton Heights, New South Wales, Australia
- Ordensklinikum Linz GmbH / Elisabethinen, Linz, Austria
- AZ Sint-Jan Brugge-Oostende av, Bruges, Belgium
- Canada (4):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Southlake Regional Health Centre, Newmarket, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec (IUCPQ), Québec, Quebec
- CMC - Clinique Ambroise Paré, Neuilly-sur-Seine, France
- Japan (4):
  - Hirosaki University Hospital, Hirosaki, Aomori
  - University of Fukui Hospital, Yoshida-gun, Fukui
  - Tokyo Medical and Dental University, Medical Hospital, Bunkyō-Ku, Tokyo
  - Jikei University, Minato-Ku, Tokyo
- St. Antonius Ziekenhuis, Nieuwegein, Netherlands
- Hospital General Universitario Gregorio Marañón, Madrid, Spain

REFERENCES:
- [Result] Verma A, Haines DE, Boersma LV, Sood N, Natale A, Marchlinski FE, Calkins H, Sanders P, Packer DL, Kuck KH, Hindricks G, Onal B, Cerkvenik J, Tada H, DeLurgio DB; PULSED AF Investigators. Pulsed Field Ablation for the Treatment of Atrial Fibrillation: PULSED AF Pivotal Trial. Circulation. 2023 May 9;147(19):1422-1432. doi: 10.1161/CIRCULATIONAHA.123.063988. Epub 2023 Mar 6. PMID 36877118
- [Result] Verma A, Boersma L, Haines DE, Natale A, Marchlinski FE, Sanders P, Calkins H, Packer DL, Hummel J, Onal B, Rosen S, Kuck KH, Hindricks G, Wilsmore B. First-in-Human Experience and Acute Procedural Outcomes Using a Novel Pulsed Field Ablation System: The PULSED AF Pilot Trial. Circ Arrhythm Electrophysiol. 2022 Jan;15(1):e010168. doi: 10.1161/CIRCEP.121.010168. Epub 2021 Dec 29. PMID 34964367
- [Derived] Yamane T, Sasano T, Tomita H, Aoyama D, Miyazaki S, Takigawa M, Kimura M, Itoh T, Yamashita S, Selma JM, Cerkvenik J, Verma A, Tada H; PULSED AF Investigators. Safety, efficacy, and quality of life outcomes of pulsed field ablation in Japanese patients with atrial fibrillation: results from the PULSED AF trial. J Interv Card Electrophysiol. 2025 Jan;68(1):149-157. doi: 10.1007/s10840-024-01912-w. Epub 2024 Sep 7. PMID 39243306
- [Derived] Verma A, Haines DE, Boersma LV, Sood N, Natale A, Marchlinski FE, Calkins H, Sanders P, Packer DL, Kuck KH, Hindricks G, Tada H, Hoyt RH, Irwin JM, Andrade J, Cerkvenik J, Selma J, DeLurgio DB; PULSED AF Investigators. Influence of monitoring and atrial arrhythmia burden on quality of life and health care utilization in patients undergoing pulsed field ablation: A secondary analysis of the PULSED AF trial. Heart Rhythm. 2023 Sep;20(9):1238-1245. doi: 10.1016/j.hrthm.2023.05.018. Epub 2023 May 19. PMID 37211146

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pilot | Pivotal - Roll-In | Pivotal - Paroxysmal AF | Pivotal - Persistent AF
Started | 38 | 60 | 164 | 159
Had Ablation Procedure | 38 | 60 | 150 | 150
Completed | 35 | 57 | 146 | 141
Not Completed | 3 | 3 | 18 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pilot | Pivotal - Roll-In | Pivotal - Paroxysmal AF | Pivotal - Persistent AF | Total
Number analyzed (Participants) | 38 | 60 | 164 | 159 | 421
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 25 | 82 | 66 | 193
  >=65 years | 18 | 35 | 82 | 93 | 228
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (11.3) | 66.7 (8.7) | 63.1 (10.4) | 65.9 (8.9) | 64.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 61 | 38 | 132
  Male | 20 | 45 | 103 | 121 | 289
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 9 | 21 | 16 | 47
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 1 | 0 | 1 | 1 | 3
  White | 34 | 45 | 121 | 128 | 328
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 6 | 20 | 14 | 42
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 5 | 7 | 5 | 25
  Austria | 0 | 1 | 0 | 6 | 7
  Netherlands | 4 | 0 | 7 | 0 | 11
  Belgium | 0 | 1 | 1 | 3 | 5
  United States | 21 | 43 | 126 | 121 | 311
  Japan | 0 | 8 | 20 | 16 | 44
  Australia | 5 | 0 | 3 | 2 | 10
  France | 0 | 1 | 0 | 2 | 3
  Spain | 0 | 1 | 0 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Safety: Number of Participants With at Least One Primary Safety Event
Description: Primary safety events are:
  Within 6 months post-ablation:
  * Pulmonary vein stenosis (≥70% diameter reduction)
  * Phrenic nerve injury/diaphragmatic paralysis (ongoing at 6 months)
  * Atrioesophageal fistula
  Within 30 days of ablation procedure:
  * Cardiac tamponade/perforation
  * Cerebrovascular accident
  * Major bleeding requiring transfusion
  * Myocardial infarction
  * Pericarditis requiring intervention
  * Transient ischemic attack
  * Vagal nerve injury resulting in esophageal dysmotility or gastroparesis
  * Vascular access complications requiring intervention
  * Systemic/pulmonary embolism requiring intervention
  * Pulmonary edema
  * Death
  * Any PulseSelect PFA System-related or PFA procedure-related cardiovascular and/or pulmonary adverse event that prolongs or requires hospitalization for more than 48 hours (excluding recurrent AF/AFL/AT)
Time Frame: up to 6 months
Population: Non roll-in pivotal patients that had a Pulsed Field Ablation procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pivotal - Paroxysmal AF | Pivotal - Persistent AF
Number analyzed (Participants) | 150 | 150
Participants | 1 | 1

2. Primary Outcome: Effectiveness: Number of Participants With Treatment Success.
Description: Treatment success is defined as freedom from treatment failure. The study requires 24-hour Holter monitoring at 6 and 12 months in addition to weekly and symptomatic patient activated ambulatory monitoring transmissions through 12 months, and 12-lead ECGs at all follow up visits. Treatment failure is defined as any of the following components:
  * Acute procedural failure
  * Documented AF/AT/AFL on Holter/patient activated ambulatory monitoring/12-lead ECG after the 90-day post-ablation blanking period.
  * Any subsequent AF surgery or ablation in the left atrium, except for one repeat PVI ablation using PFA within the 90-day blanking period.
  * Direct current cardioversion for atrial tachyarrhythmia recurrences after the 90-day blanking period.
  * Class I or III antiarrhythmic drug (AAD) dose increase from the historic maximum ineffective dose (prior to the ablation procedure) or initiation of a new Class I or III AAD after the 90-day blanking period.
Time Frame: up to 12 months
Population: Non roll-in pivotal patients that had a Pulsed Field Ablation procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pivotal - Paroxysmal AF | Pivotal - Persistent AF
Number analyzed (Participants) | 150 | 150
Participants | 100 | 83

3. Secondary Outcome: Quality of Life - Change in EQ-5D Score
Description: Change in EQ-5D score (12-month score - baseline score). The Euroqol EQ-5D questionnaire (5L version) is a standardized instrument for measuring general health status. The Euroqol EQ-5D questionnaire (which consists of a 5-question survey and a visual analog scale) has a composite score based on the 5-question survey that ranges from 0 (least healthy) to 1 (most healthy).
Time Frame: Baseline to 12 months post-ablation
Population: All participants who completed the EQ-5D questionnaire at baseline and 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pivotal - Paroxysmal AF | Pivotal - Persistent AF
Number analyzed (Participants) | 144 | 140
units on a scale | 0.05 [0.02 to 0.08] | 0.06 [0.04 to 0.09]

4. Secondary Outcome: Quality of Life - Change in AFEQT Score
Description: Change in AFEQT score (12-month score - baseline score). The AFEQT questionnaire is an atrial fibrillation (AF) specific health-related quality of life questionnaire to assess the impact of AF on a subject's life. The overall score ranges from 0 - 100, with 0 corresponding to complete disability and 100 corresponding to no disability
Time Frame: Baseline to 12 months post-ablation
Population: All participants who completed the AFEQT questionnaire at baseline and 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pivotal - Paroxysmal AF | Pivotal - Persistent AF
Number analyzed (Participants) | 144 | 140
units on a scale | 29.4 [25.8 to 33.1] | 29.0 [25.5 to 32.5]

5. Other Pre Specified Outcome: Pilot Phase Safety: Number of Participants With a PFA System-related and PFA Procedure-related Serious Adverse Event (SAE) Within 30 Days Post-ablation.
Description: Serious adverse events that count toward the endpoint are:
  Pulmonary vein stenosis (>70% diameter reduction) Atrioesophageal fistula Cardiac tamponade/perforation Cerebrovascular accident Major bleeding requiring transfusion Myocardial infarction Pericarditis requiring intervention Transient ischemic attack Vagal nerve injury resulting in esophageal dysmotility or gastroparesis Vascular access complications requiring intervention Systemic/pulmonary embolism requiring intervention Pulmonary edema Death
Time Frame: 30 days
Population: Pilot patients
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot
Number analyzed (Participants) | 38
Participants | 0

6. Other Pre Specified Outcome: Pilot Phase Effectiveness: Number of Participants With Acute Procedural Success of PVI Ablation With the PFA System.
Description: Acute procedural failure is defined as the occurrence of any of the following:
  1. Inability to isolate all accessible targeted pulmonary veins (assessed for entrance block and, where assessable, exit block) during the index ablation procedure.
  2. Ablation using a non-study device in the left atrium.
  Acute procedural success is the opposite of acute procedural failure.
Time Frame: Acute (day of procedure)
Population: Pilot patients
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot
Number analyzed (Participants) | 38
Participants | 38

ADVERSE EVENTS:
Time Frame: Study enrollment to 12 months post-ablation
Description: All adverse events were collected.
  Serious adverse event:
  Adverse event that
  1. led to death,
  2. led to serious deterioration in the health as defined by one or more of the following:
     1. a life-threatening illness or injury, or
     2. a permanent impairment of a body structure, including chronic disease, or
     3. in-patient or prolonged hospitalization, or
     4. medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment
Arm/Group | Pilot | Pivotal - Roll-In | Pivotal - Paroxysmal AF | Pivotal - Persistent AF
All-Cause Mortality (participants affected / at risk) | 1/38 | 1/60 | 1/164 | 1/159
Serious Adverse Events (participants affected / at risk) | 13/38 | 20/60 | 38/164 | 56/159
Other Adverse Events (participants affected / at risk) | 19/38 | 17/60 | 39/164 | 53/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilot (N=38) | Pivotal - Roll-In (N=60) | Pivotal - Paroxysmal AF (N=164) | Pivotal - Persistent AF (N=159)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 8 (10) | 7 (7) | 14 (14) | 27 (29)
Atrial flutter (Cardiac disorders) | 1 (1) | 5 (5) | 6 (6) | 6 (6)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Retention cyst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Diabetic gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphatic duct injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilot (N=38) | Pivotal - Roll-In (N=60) | Pivotal - Paroxysmal AF (N=164) | Pivotal - Persistent AF (N=159)
Atrial fibrillation (Cardiac disorders) | 7 (15) | 8 (10) | 17 (20) | 30 (37)
Atrial flutter (Cardiac disorders) | 3 (4) | 3 (3) | 9 (12) | 11 (13)
Atrial tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Palpitations (Eye disorders) | 5 (6) | 0 (0) | 3 (3) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 4 (4)
Ventricular extrasystoles (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Chest pain (General disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 11 (11) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan: version 7 (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/01/NCT04198701/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: version 6 (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/01/NCT04198701/Prot_SAP_001.pdf
  • Study Protocol and Statistical Analysis Plan: version 3 (2020-01-19): https://cdn.clinicaltrials.gov/large-docs/01/NCT04198701/Prot_SAP_002.pdf
  • Study Protocol and Statistical Analysis Plan: version 2 (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT04198701/Prot_SAP_003.pdf